CLINICAL TRIAL: NCT04008550
Title: Prognostic Impact of the Evolution of Pulmonary Arterial Hypertension 3 Months After Transcatheter Aortic Valve Implantation
Brief Title: Prognostic Impact of the Evolution of PAH 3 Months After TAVI (HTP-TAVI)
Acronym: HTP-TAVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Delay in enrolment (24% at 1 year)
  * Lower than estimated prevalence of PAH (15% instead of 50%)
  * Refusal of patients with PAH to participate
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/093/HP
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Aortic Valve Stenosis; Pulmonary Hypertension
Keywords: TAVI (Transcatheter Aortic Valve Implantation); Aortic Stenosis; Pulmonary Arterial Hypertension; Right Heart Catheterization
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Pulmonary Arterial Hypertension before TAVI (No Intervention): No intervention has been done in this group of patients.
- Pulmonary Arterial Hypertension before TAVI (Other): In this group, a right heart catheterization is done 3 months after TAVI in order to evaluate PAH (persistence or regression).
  Interventions: Procedure: Right Heart Catheterization

INTERVENTIONS:
Procedure: Right Heart Catheterization — A right heart catheterization will be done in patients with PAH before TAVI (3 months after TAVI)
  Arms: Pulmonary Arterial Hypertension before TAVI

SUMMARY:
Aortic stenosis (AS) is the most frequent valvulopathy in Western countries. The prevalence of AS is constantly increasing due to the aging of the population. Several studies have shown that pulmonary arterial hypertension (PAH) was common in AS patients referred for TAVI and that it was an independent predictor of mortality after TAVI.

Currently, there is no data in the literature regarding the evolution and prognosis value of PAH measured using right heart catheterization (reference method). PAH could either regress after TAVI or continue to progress despite the treatment of valvulopathy, resulting in a refractory right heart failure that can lead to death.

The hypothesis of this study is that patients with PAH before TAVI procedure and at the 3-month follow-up visit (PAH persistence) have an increased risk of cardiovascular mortality compared to patients with no PAH at 3 months or having a significant reduction of their PAH (PAH regression).

The aim of the study is to evaluate the prognostic impact of the evolution of PAH after TAVI in 424 patients using right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis
* Indication of TAVI

Exclusion Criteria:

* Contra-indication of right heart catheterization
* Pregnancy
* Persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Hospitalization for heart failure or death any cause (composite endpoint) | Up to 24 months
  Time before the first event (hospitalization or death any cause)

SECONDARY OUTCOMES:
Post-operative evolution of the PAH, according to the type of pre-operative PAH | Year 2
  PAPm (mean pulmonary arterial pressure) measurement
Prevalence of pre-TAVI PAH | Year 0
  In percent and according to the type of PAH (pre-TAVI)
Hospital-free survival for heart failure among the 3 types of PAH (pre-TAVI) | Year 2
  Occurrence of clinical events
Prognosis (survival without hospitalization for heart failure) of subjects whose PAH corrected post-TAVI to those who had no pre-TAVI PAH | Month 3
  Occurrence of clinical events
Concordance between the PAH measurement techniques: echocardiography and right heart catheterization | Month 3
  PAPm (mean pulmonary arterial pressure) measurement (Echocardiography or right heart catheterization)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Durand, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France